CLINICAL TRIAL: NCT01324219
Title: Changing Talk to Reduce Resistiveness to Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 12146
Record Dates: First submitted 2011-03-16; First posted 2011-03-28 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Dementia
Keywords: nursing staff; residents
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Staff (Active Comparator)
  Interventions: Behavioral: Staff
- Resident (Experimental)
  Interventions: Behavioral: Resident

INTERVENTIONS:
Behavioral: Staff — Your participation will involve participating in video recordings of nursing care for a participating resident for 2-hour periods on 8 to 10 days. Communication training will be provided to staff in participating nursing homes during paid work hours regardless of their participation in the video recordings. The nursing home you work in may be randomly selected to receive the communication training at the start of the study or after a 3-month delay.
  Arms: Staff
Behavioral: Resident — Your participation will involve participating in video recordings of nursing care for 2-hour periods on 8 to 10. Communication training will be provided to staff in participating facilities during paid work hours regardless of their participation in the video recordings. Your nursing home may be randomly selected to receive the communication training at the start of the study or after a 3-month delay.
  Arms: Resident

SUMMARY:
The investigators are interested in reducing problem behaviors of nursing home residents with dementia that make providing care difficult. The investigators call these behaviors resistiveness to care. Previous research has found that resistiveness to care occurs more frequently when staff use certain types of communication. An inservice program will be provided to all nursing staff in your nursing home to teach staff about communication practices to reduce resistiveness to care. The research study will see whether changing communication will reduce resident resistiveness to care. If effective, the communication training may then be used to improve care in other facilities.

By doing this study, researchers hope to learn if changing communication practices will reduce resistiveness to care in nursing home residents with dementia.

ELIGIBILITY:
Staff:Inclusion criteria for CNAs are:

* age 18 years old or greater (age of legal consent in Kansas and Missouri), signed informed consent,
* permanent employment in the NH,
* primary assignment to a specified unit,
* and English speaking
* Staff must have been assigned to care for the resident at least twice weekly in the past month (documented in NH staffing records). This will assure that staff-resident dyads have established relationships and will control effects of variability in contact between dyads during days when data are not being collected.

Resident inclusion criteria are:

* a diagnosis of Alzheimer's disease or related dementia documented in their medical records,
* documentation of daily RTC over the past week,
* and ability to hear staff communication (from the most recent MDS).

Exclusion criteria for CNAs include:

* non-English speaking,
* temporary employment, -and age under 18 years.
* If more than one CNA volunteers as a partner for a participating resident, a random selection will be made to determine which CNA will participate. Small variations in contact between staff and residents in dyads are anticipated due to PMMA policies for consistent CNA assignment to neighborhoods. Therefore dyads will have repeated contacts.

Exclusion criteria for residents include:

* diagnosis with Huntington's disease,
* alcohol-related dementias,
* schizophrenia,
* manic-depressive disorder,
* deafness,
* and mental retardation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the effects of the nursing staff communication - change in frequency and duration of resident Resistiveness to Care behaviors. | up to 6 months
  Test the effects of the CHAnging Talk (CHAT) nursing staff communication intervention on reducing the frequency and duration of resident Resistiveness to Care (RTC) behaviors.

SECONDARY OUTCOMES:
Calculate the costs of nursing staff communication system | up to 6 months
  Calculate the costs of CHAT using traditional methods and assess its cost-effectiveness with innovative Data Envelopment Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Williams, RN, PhD, APRN, FNP-BC, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Liu W, Perkhounkova Y, Williams K, Batchelor M, Hein M. Mealtime nonverbal behaviors in nursing home staff and residents with dementia: Behavioral analyses of videotaped observations. Geriatr Nurs. 2022 Mar-Apr;44:112-124. doi: 10.1016/j.gerinurse.2022.01.009. Epub 2022 Feb 4. PMID 35131660
- [Derived] Liu W, Batchelor M, Williams K. Development and Psychometric Testing of the Mealtime Engagement Scale in Direct Care Providers of Nursing Home Residents With Dementia. Gerontologist. 2021 Nov 15;61(8):e410-e420. doi: 10.1093/geront/gnaa097. PMID 32726447
- [Derived] Jao YL, Liu W, Williams K, Chaudhury H, Parajuli J. Association between environmental stimulation and apathy in nursing home residents with dementia. Int Psychogeriatr. 2019 Aug;31(8):1109-1120. doi: 10.1017/S1041610219000589. PMID 31241031
- [Derived] Williams KN, Perkhounkova Y, Herman R, Bossen A. A Communication Intervention to Reduce Resistiveness in Dementia Care: A Cluster Randomized Controlled Trial. Gerontologist. 2017 Aug 1;57(4):707-718. doi: 10.1093/geront/gnw047. PMID 27048705